CLINICAL TRIAL: NCT07246967
Title: An International Multicenter Study on the Antimicrobial Prophylaxis Strategy for Flexible Ureteroscopic Lithotripsy Combined With a Flexible Negative Pressure Suction Sheath
Brief Title: Antibiotic Prophylaxis for Ureteroscopy With a Negative Pressure Suction Sheath
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yi Shao, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT2025-208
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Urolithiasis; Antibiotics
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Undergo flexible ureteroscopic lithotripsy and stone clearance with a flexible negative-pressure sheath without the use of any prophylactic antimicrobials; postoperatively, therapeutic antimicrobials will be initiated only for patients who develop signs or symptoms of infection.
  Interventions: Drug: not use any prophylactic antimicrobials
- Group 2 (Active Comparator): Receive a single dose of intravenous prophylactic antimicrobials (e.g., a second-generation cephalosporin or levofloxacin) 30-60 minutes before surgery, followed by the same standardized flexible negative-pressure sheath ureteroscopic surgery.
  Interventions: Drug: use prophylactic antimicrobials

INTERVENTIONS:
Drug: not use any prophylactic antimicrobials — The experimental group will undergo surgery without the use of any prophylactic antimicrobials; therapeutic antimicrobials will only be administered postoperatively to patients who develop signs or symptoms of infection. The control group will receive a single dose of intravenous prophylactic antimicrobials 30-60 minutes before surgery, followed by the same standardized surgical procedure.
  Other Names: without the use of any antimicrobial drugs for prophylaxis
  Arms: Group 1
Drug: use prophylactic antimicrobials — Receive a single dose of intravenous prophylactic antimicrobials (e.g., a second-generation cephalosporin or levofloxacin) 30-60 minutes before surgery, followed by the same standardized flexible negative-pressure sheath ureteroscopic surgery.
  Other Names: apply antimicrobial drugs for prophylaxis
  Arms: Group 2

SUMMARY:
This study, as a prospective, randomized, controlled, non-inferiority, international multicenter clinical trial, aims to evaluate whether a strategy of no antimicrobial prophylaxis is non-inferior to the traditional single-dose prophylaxis regimen in patients with a low risk of infection undergoing single-use flexible ureteroscopic lithotripsy combined with a flexible negative-pressure suction sheath. It is anticipated that this will have a substantial impact on infection prevention strategies in urological surgery.

DETAILED DESCRIPTION:
This study, as a prospective, randomized, controlled, non-inferiority, international multicenter clinical trial, aims to evaluate whether a strategy of no antimicrobial prophylaxis is non-inferior to the traditional single-dose prophylaxis regimen in patients with a low risk of infection undergoing single-use flexible ureteroscopic lithotripsy combined with a flexible negative-pressure suction sheath. It is anticipated that this will have a substantial impact on infection prevention strategies in urological surgery.

This trial is an international, multicenter, prospective, randomized controlled trial. The participating centers are: Shanghai General Hospital (lead institution), Shanghai Xinhua Hospital, Weifang Traditional Chinese Medicine Hospital, School of Medicine, Mulawarman University Abdul Wahab Sjahranie Hospital (Indonesia), and Hospital Raja Perempuan Zainab II (Malaysia).

This trial will employ a non-inferiority design and a central randomization system to allocate eligible subjects in a 1:1 ratio to either the experimental group (no prophylactic antimicrobials) or the control group (single-dose antimicrobial prophylaxis). Stratification factors will include the participating center and stone size, with subjects stratified by the longest stone diameter: ≤1.5cm and >1.5cm but ≤2cm.

All surgeries will be performed by surgeons with experience of ≥50 cases of flexible negative-pressure sheath procedures, using a standardized surgical record form to document key operational parameters (e.g., sheath model, negative pressure settings, operative time, irrigation volume, etc.). Prior to study initiation, all centers will undergo standardized surgical video training and simulated operational assessments to ensure technical consistency.

The surgery will follow standardized technical parameters: a F10/12, F11/13, or F12/14 flexible negative-pressure sheath will be selected based on the patient's ureteral conditions; the central negative pressure will be set to 0.02-0.04MPa; the irrigation flow rate will be 50-150 ml/min, adjusted to the minimum rate that both maintains collecting system filling and ensures low intrarenal pressure; and the lithotripsy will employ a 'simultaneous fragmentation and suction for in-situ stone clearance' strategy.

The study subjects will be patients with a low risk of infection (defined as no preoperative symptoms of infection such as chills and fever, a negative urine culture, and a stone size ≤2cm) from multiple centers who are scheduled to undergo single-use flexible ureteroscopic lithotripsy combined with a flexible negative-pressure suction sheath. They will be allocated in a 1:1 ratio to the experimental group or the control group. The experimental group will undergo surgery without the use of any prophylactic antimicrobials; therapeutic antimicrobials will only be administered postoperatively to patients who develop signs or symptoms of infection. The control group will receive a single dose of intravenous prophylactic antimicrobials 30-60 minutes before surgery, followed by the same standardized surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Diagnosed by CT with renal and/or upper ureteral stones, with the longest stone diameter being ≤2cm.
3. Scheduled to undergo fURS lithotripsy.
4. No preoperative symptoms of infection such as chills and fever, and the most recent preoperative urine culture is negative.
5. No immunosuppressive status and no urinary flow obstruction caused by anatomical abnormalities.
6. No use of long-acting antimicrobial agents within 7 days prior to surgery, and no use of intermediate or short-acting antimicrobial agents within 72 hours prior to surgery.
7. Has signed and dated an informed consent form, indicating that the patient or their legal representative has been fully informed about the study-related information and has agreed to participate.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Allergy to the investigational drug(s).
3. Participation in other clinical trials within 30 days.
4. Presence of other active infection foci requiring antimicrobial treatment.
5. Concomitant severe systemic diseases, such as cardiac or pulmonary disease, malignant tumors, and immunodeficiency states.
6. Congenital malformations of the urinary tract.
7. History of kidney transplantation or urinary diversion surgery.
8. Unable to provide samples or complete follow-up according to the study protocol.
9. Unable to provide informed consent.
10. Inability to achieve complete placement of the flexible negative-pressure suction sheath.
11. Any other conditions that the investigator deems unsuitable for participation in this study.
12. History of diabetes mellitus, immunocompromised.
13. Renal insufficiency, neurogenic bladder.
14. Recent preoperative history of stone-related fever.
15. Long-term indwelling urinary drainage tube.
16. Urine white blood cells >5/HPF (High Power Field) or positive for urine nitrites.
17. Large stone burden (e.g., staghorn calculus) or moderate to severe hydronephrosis.
18. Imaging findings showing turbid urine in the renal pelvis where pyonephrosis or infectious stones cannot be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of Systemic Inflammatory Response Syndrome (SIRS) within 72 hours postoperatively | within 72 hours postoperatively
  To reduce the influence of subjective factors and to more comprehensively reflect the systemic inflammatory state, the primary endpoint is the incidence of Systemic Inflammatory Response Syndrome (SIRS) within 72 hours postoperatively, defined as meeting at least two of the following criteria:
  Body temperature >38°C or <36°C Heart rate >90 beats/minute Respiratory rate >20 breaths/minute or PaCO2 <32 mmHg White blood cell count >12×10⁹/L or <4×10⁹/L, or >10% immature neutrophils

CONTACTS AND LOCATIONS:
Overall Officials: Yi Shao, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
After the trial is completed, it is shared on the network platform: China Clinical trial Registration Center; website: http://www.chictr.org.cn
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the trial is completed
URL: http://www.chictr.org.cn